CLINICAL TRIAL: NCT02155504
Title: A Phase 1, Single Ascending Oral Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP3700 in Healthy Male Subjects, Including a Drug-drug Interaction Part With Itraconazole
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP3700 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3700-CL-0001; 2013-005018-36 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-06-04 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers; Pharmacokinetics of ASP3700
Keywords: Healthy volunteers; Pharmacokinetics; ASP3700; Itraconazole; Drug-drug interaction
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP3700 single ascending dose cohort (Experimental): Part 1
  Interventions: Drug: ASP3700
- Placebo single ascending dose cohort (Placebo Comparator): Part 1
  Interventions: Drug: Placebo
- ASP3700 alone (Experimental): Part 2
  Interventions: Drug: ASP3700
- ASP3700 and itraconazole (Active Comparator): Part 2
  Interventions: Drug: ASP3700; Drug: itraconazole

INTERVENTIONS:
Drug: ASP3700 — oral
  Arms: ASP3700 alone; ASP3700 and itraconazole; ASP3700 single ascending dose cohort
Drug: itraconazole — oral
  Arms: ASP3700 and itraconazole
Drug: Placebo — oral
  Arms: Placebo single ascending dose cohort

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of single ascending oral doses of ASP3700 in healthy male subjects. This study will also explore the effect of itraconazole (another drug) on the PK of ASP3700, as well as to evaluate the safety and tolerability of ASP3700 alone and in combination with itraconazole in healthy male subjects.

DETAILED DESCRIPTION:
This study consists of 2 parts: Part 1 is a single ascending dose study where subjects will receive either ASP3700 or matching placebo; Part 2 is a drug-drug interaction (DDI) open-label, crossover study comprised of 1 sequence with 2 investigational periods where subjects will receive ASP3700 alone and in combination with itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 - 30.0 kg/m2. The subject weighs at least 50 kg.
* Subject and his female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continue throughout the clinical study period and for 90 days after the final study drug administration.
* Subject must not donate sperm starting at screening and throughout the clinical study period and for 90 days after the final study drug administration.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to ASP3700 (parts 1 and 2) or itraconazole (part 2 only) or significant adverse reactions to historical cannabinoid use or any components of the formulations used.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma-glutamyl transaminase, total bilirubin [TBL]) above the upper limit of normal (ULN). In such a case the assessment may be repeated once (upon admission to the clinical unit).
* Subject has a history of a suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 3 months or who are at significant risk to commit suicide, as judged by the Investigator using the C-SSRS (a level of 4 or 5) at screening or upon admission to the clinical unit.
* Subject has any clinically significant abnormality following the Investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or upon admission to the clinical unit.
* Subject has a pulse rate < 40 or > 90 beats per minute; mean SBP > 140 mmHg; mean DBP > 90 mmHg (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse rate will be measured automatically) upon admission to the clinical unit.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) interval > 430 ms at day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit.
* Subject has a history of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit.
* Subject has consumed grapefruit, grapefruit-containing products or Seville orange-containing products within 72 hours prior to admission to the clinical unit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events (Part 1) | up to end of study visit (up to 16 days)
Safety as assessed by vital signs (Part 1) | up to end of study visit (up to 16 days)
Safety as assessed by laboratory tests (Part 1) | up to end of study visit (up to 16 days)
  Laboratory tests includes the measurement of sex-hormone related biomarkers and exploratory renal biomarkers.
Safety as assessed by electrocardiogram (ECG) measurements (Part 1) | up to end of study visit (up to 16 days)
  ECG measurements include routine 12-lead ECG, continuous cardiac monitoring (Holter ECG) and real-time cardiac monitoring (ECG telemetry)
Safety as assessed by Bond and Lader VAS (Part 1) | Up to Day 2
  visual analogue scale (VAS)
Safety as assessed by C-SSRS (Part 1) | Up to end of study visit (up to 16 days)
  Columbia - Suicide Severity Rating Scale (C-SSRS)
Safety as assessed by ARCI-49 (Part 1) | Up to Day 2
  Addiction Research Center Inventory (ARCI)-49 (49-item)
Pharmacokinetic parameter of itraconazole (plasma): Ctrough (Part 2) | Days 3-13
  Concentration immediately prior to dosing at multiple dosing
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): AUCinf (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Area under the concentration-time curve from time of dosing extrapolated to time infinity (AUCinf)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): AUCinf (%extrap) (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Percentage of AUCinf due to extrapolation from tlast to time infinity (AUCinf [%extrap])
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): AUClast (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): Cmax (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Maximum concentration (Cmax)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma):λz (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Terminal elimination rate constant (λz)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): MRT (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Mean residence time (MRT)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): tlag (Part 2) | Day 1 (period 1 and 2)
  Time prior to the time corresponding to the first measurable (nonzero) concentration (tlag)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): tmax (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Time of maximum concentration (tmax)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): t1/2 (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Terminal elimination half-life (t1/2)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (plasma): Vz/F (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (urine): Aelast (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Cumulative amount of study drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (urine): Aeinf (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (urine): Aelast% (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Percentage of study drug excreted into urine from the time of dosing up to the collection time of the last measurable concentration (Aelast%)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (urine): Aeinf% (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Percentage of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf%)
Pharmacokinetic parameter of ASP3700 with and without itraconazole (urine): CLR (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2)
  Renal clearance (CLR)
Safety as assessed by orthostatic evaluation (or blood pressure change in orthostatic challenge test) (Part 1) | Up to Day 7

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP3700: AUCinf, AUCinf(%extrap), AUClast, Cmax, CL/F, λz, MRT, tlag, tmax, t½, Vz/F (plasma) (Part 1) | up to Day 7
Title: Composite of pharmacokinetics of ASP3700: Aelast, Aeinf, Aelast%, Aeinf%, CLR (urine) (Part 1) | up to Day 7
Safety as assessed by adverse events, vital signs, orthostatic evaluation, laboratory tests, ECG measurements, C-SSRS, Bond & Lader VAS, ARCI-49 (Part 2) | Days 1-7 (period 1) and Days 1-13 (period 2) and at end of study visit (up to 22 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, United Kingdom